CLINICAL TRIAL: NCT00482547
Title: Study of a Urethral Catheter Coated With Eluting Silver Salts
Brief Title: Study of a Urethral Catheter Coated With Eluting Silver Salts (SUCCESS)
Acronym: SUCCESS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated for futility reasons.
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMD-6003
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Results first posted 2010-01-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Catheterization
Keywords: urinary tract infection; urinary catheter
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silver-coated catheter (Experimental): Bard Hydrogel Silver Salts Coated Latex Urinary Catheter System
  Interventions: Device: Hydrogel Silver Salts Coated Latex Urinary Catheter System
- Silicone-coated catheter (Placebo Comparator): Bard silicone elastomer coated latex catheter system
  Interventions: Device: Bard silicone elastomer coated latex catheter system

INTERVENTIONS:
Device: Hydrogel Silver Salts Coated Latex Urinary Catheter System — Silver-coated catheter
  Other Names: AgSC arm
  Arms: Silver-coated catheter
Device: Bard silicone elastomer coated latex catheter system — Silicone-coated catheter
  Other Names: SiCS arm
  Arms: Silicone-coated catheter

SUMMARY:
Urinary catheters are often needed in hospital patients, but their use can increase the chance that a catheter associated urinary tract infection (called a CAUTI) may occur. This study will try to determine if patients who get a new silver coated catheter will have slower to time to development of a CAUTI compared to patients who get an uncoated catheter.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled pivotal study designed to compare the time to occurrence and incidence of CAUTI in subjects catheterized with a new hydrogel-silver salts latex catheter (test) to those of subjects catheterized with a silicone elastomer-coated latex catheter (control).

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 18 years of age
* life expectancy of 3 months or more
* expected to require a urinary catheter for at least 48 hours

Exclusion Criteria:

* recent urinary tract surgery or instrumentation
* presence of a urinary tract device
* concurrent genitourinary tract infection
* recent indwelling urinary catheter
* requires use of a non-study urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1188 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rupp, MD, Principal Investigator — University of Nebraska
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty Investigators at 20 Investigative Sites enrolled a total of 1188 study subjects between June 28, 2007 and June 23, 2008.
Pre-assignment Details: Subjects judged by site personnel to require a urinary catheter for at least 48-72 hours were screened against the study inclusion/exclusion criteria. Those subjects meeting these criteria were offered participation in the study.
Groups:
- Silver-coated Catheter: Bard® Hydrogel Silver Salts Coated Latex Urinary Catheter
- Silicone-coated Catheter: silicone elastomer-coated latex catheter
Period: Overall Study
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Started | 599 (599 subjects were enrolled in the silver-coated catheter group.) | 589 (589 subjects were enrolled in the silicone-coated catheter group.)
Successful Catheterization | 565 (Out of the 599 AgCS subjects 565 (94.3%) had a successful catheterization.) | 568 (Out of the 589 SiCS catheter subjects 568 (96.4%) had a successful catheterization.)
48 Hour Evaluation | 426 (426 went on to be included in the Silver-coated 48 hour efficacy evaluable population.) | 428 (428 went on to be included in the Silicone-coated 48 hour efficacy evaluable population.)
Completed | 426 | 428
Not Completed | 173 | 161

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter | Total
Number analyzed (Participants) | 599 | 589 | 1188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 302 | 287 | 589
  >=65 years | 297 | 302 | 599
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (15.9) | 64.3 (14.5) | 64.0 (15.2)
Gender [Count of Participants; unit: Participants]
  Female | 341 | 332 | 673
  Male | 258 | 257 | 515
Region of Enrollment [Number; unit: participants]
  United States | 599 | 589 | 1188.0

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With a bUTI After Catheterization for >= 48 Hours
Description: The percentage of bUTI was calculated as the rate of new occurrence of bUTI in subjects of both study groups who had been catheterized with a study catheter for >= 48 hours and who did not have evidence of bUTI at the time of study catheter insertion.
Time Frame: >=48 hours to 10 days
Population: Efficacy Evaluable (48) population: ITT subjects who were catheterized with a study catheter for ≥ 48 hours and who did not have a bUTI in the baseline urine sample obtained at the time of catheter insertion.
Measure: Number; unit: Percentage of Participants with a bUTI
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 426 | 428
Percentage of Participants with a bUTI | 13.4 | 17.8

2. Primary Outcome: Time to Occurrence of Bacteriuric Urinary Tract Infection (bUTI) in Subjects Catheterized for >= 48 Hours
Description: Time to occurrence of bUTI in subjects of both study groups who were catheterized with a study catheter for >= 48 hours and who had evidence of bUTI after study catheter insertion. Subjects who did not have a bUTI are not included in the median calculation, so the median only includes data from non-censored observations.
Time Frame: >=48 hours to 10 days
Population: Efficacy Evaluable (48) population: Intent-to-treat (ITT) subjects who were catheterized with a study catheter for ≥ 48 hours and who developed a bUTI after catheter insertion.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 57 | 76
Days | 2.10 (1.99) | 2.06 (2.32)

3. Secondary Outcome: Time to Occurence of Symptomatic Urinary Tract Infection (sUTI) in Subjects Catheterized for >= 48 Hours
Description: The time to occurrence of sUTI was measured as the time between catheter insertion and when the criteria for sUTI was met, up to 10 days after catheterization plus 48 hours after catheter removal. Subjects who did not have a sUTI are not included in the median calculation, so the median only includes data from non-censored observations.
Time Frame: >= 48 hours to 10 days
Population: Efficacy Evaluable (48) population: ITT subjects who were catheterized with a study catheter for ≥ 48 hours and who developed a sUTI after catheter insertion.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 37 | 38
Days | 1.23 (1.75) | 1.62 (1.48)

4. Secondary Outcome: Time to Occurence of bUTI in Subjects Catheterized for >= 24 Hours
Description: Time to occurrence of bUTI in subjects of both study groups who were catheterized with a study catheter for >= 24 hours and developed a bUTI at after catheter insertion. Subjects who did not have a bUTI are not included in the median calculation, so the median only includes data from non-censored observations.
Time Frame: >= 24 hours to 10 days
Population: Efficacy Evaluable (24) population: ITT subjects who were catheterized with a study catheter for ≥ 24 hours and who developed a bUTI after catheter insertion.
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 61 | 78
Days | 2.03 (1.98) | 2.04 (2.31)

5. Secondary Outcome: Time to Occurance of sUTI in Subjects Catheterized for >= 24 Hours
Description: as for outcome 3
Time Frame: >= 24 hours to 10 days
Population: as for outcome 4
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 39 | 39
Days | 1.1039 (1.73) | 1.40 (1.47)

6. Secondary Outcome: Number of Participants With Bacteriuria at a Concentration of ≥ 10e3 < 10e5 CFU/mL
Description: The number of subjects with bacteriuria levels ≥ 10e3 < 10e5 CFU/mL who subsequently developed a bUTI or a sUTI
Time Frame: 10 days
Population: Safety population: ITT subjects who were catheterized with a study catheter. This population was used to assess tolerability and safety endpoints.
Measure: Number; unit: Participants
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 565 | 568
Participants | 38 | 35

7. Other Pre Specified Outcome: Number of Subjects With a bUTI Catheterized for >=48 Hours.
Description: bUTI occurences were counted in subjects of both study groups who had been catheterized with a study catheter for >= 48 hours and who did not have evidence of bUTI at the time of study catheter insertion.
Time Frame: From time of catheterization until 10 days post catheterization or 48 hours after catheter removal.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 426 | 428
Participants | 57 | 76

8. Other Pre Specified Outcome: Number of Subjects With a sUTI Catheterized for >=48 Hours.
Description: sUTI occurences were counted in subjects of both study groups who had been catheterized with a study catheter for >= 48 hours and who did not have evidence of bUTI at the time of study catheter insertion.
Time Frame: From time of catheterization until 10 days or 48 hours after catheter was removed
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Number analyzed (Participants) | 426 | 428
Participants | 37 | 38

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of attempted or successful catheter insertion throughout the period of catheterization with the study catheter and for a period of 48 hours following study catheter removal, or until hospital discharge.
Description: AE Definition: any undesirable clinical occurrence in a subject that is related to either the urinary tract, or systemic infection.
  All SAEs were collected, as defined in 21 CFR 803.3.
Arm/Group | Silver-coated Catheter | Silicone-coated Catheter
Serious Adverse Events (participants affected / at risk) | 47/565 | 58/568
Other Adverse Events (participants affected / at risk) | 15/565 | 29/568
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Silver-coated Catheter (N=565) | Silicone-coated Catheter (N=568)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 14
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased Bronchial Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 4
Cardiac Arrest (Cardiac disorders) | 1 | 3
Ventricular Tachycardia (Cardiac disorders) | 2 | 2
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 3
Septic Shock (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 1
Postoperative Ileus (Injury, poisoning and procedural complications) | 1 | 2
Abdominal Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 1
Reocclusion (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Acute Prerenal Failure (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Cerebellar Haemorrhage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Syncope Vasovagal (Nervous system disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 1
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Chest Pain (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 0 | 1
Blood Amylase Increased (Investigations) | 1 | 0
Blood Creatine Increased (Investigations) | 1 | 0
Lipase Increased (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Wound Drainage (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Silver-coated Catheter (N=565) | Silicone-coated Catheter (N=568)
Haematuria (Renal and urinary disorders) | 12 | 15
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 | 14

LIMITATIONS AND CAVEATS:
Sample size calculations required 1244 Efficacy Evaluable 48 subjects, only 854 Efficacy Evaluable 48 subjects were enrolled, which does not allow for a fully powered study and there is the threat of a type II error (false negative result).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days